CLINICAL TRIAL: NCT05202873
Title: Comparative Analysis of Spatiotemporal Gait Parameters in Patients With Distal Femoral Megaprosthesis and Healthy Subjects Using an Inertial Measurement Unit (IMU)
Brief Title: Analysis of Spatiotemporal Gait Parameters in Patients With Megaprosthesis.
Acronym: MP-GP
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor of the Deparment of Biomedical Sciences, Cardenal Herrera University
Other Study IDs: UNIVERSITY CARDENAL HERRERA-62
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Distal Femoral Musculoskeletal Tumors; Megaprosthesis
Keywords: Gait Analysis; Case-control study; Megaprosthesis; Orthopedic oncology; Musculoskeletal tumour; Distal femur; Inertial Measurement Unit
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with distal femoral megaprosthesis due to musculoskeletal tumor
  Interventions: Diagnostic Test: Gait analysis
- Control: Healthy subjects
  Interventions: Diagnostic Test: Gait analysis

INTERVENTIONS:
Diagnostic Test: Gait analysis — Gait assessment will be performed using a non-invasive device. It is the BTS G-sensor inertial sensor (BTS Bioengineering, Garbagnate Milanese, Italy). The spatiotemporal variables of gait will be studied from the Walk+ protocol, in which the participant navigates a 7-meter hallway six times, completing three round trips with necessary turns at each end to change direction.

SUMMARY:
The main objective of the study is to evaluate spatiotemporal parameters of gait in tumoral patients with megaprosthesis of the distal femur.

DETAILED DESCRIPTION:
Patients with distal femoral prostheses treated at La Fe Hospital in Valencia were evaluated and compared with healthy controls. A radiographic study was conducted in cases using telemetric imaging to assess the percentage of remaining bone and the long length limb discrepancy following surgical intervention. Additionally, a gait analysis was performed using the BTS device to obtain objective gait parameters. The gait assessment was conducted with a non-invasive portable device, the BTS G-sensor inertial sensor (BTS Bioengineering, Garbagnate Milanese, Italy), which was placed at the S1 level to collect spatio-temporal gait data. The data were analyzed in relation to the values in healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* Megaprosthesis of the distal femur
* Tumor cause
* Surgery at Hospital la Fe.
* Traditional stem or biological ossteointegration system
* Minimum postoperative follow-up period of 3 months

Exclusion Criteria:

* Neurological alterations prior to the intervention that affect the lower limbs or general movement.
* Patient incapable of ambulation due to progression of his/her pathology
* Patient at home with palliative treatment for advanced tumor disease
* Any ipsilateral or contralateral prosthesis.
* Infectious or traumatic cause

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent a megaprosthesis of the lower limb (distal femur) at Hospital La Fe by the orthopedic surgery and traumatology service, due to a tumor cause
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Antero-posterior acceleration symmetry index | 3 months
  This metric serves as a quantifiable measure of the symmetry exhibited in movements along the antero-posterior axis, thereby illustrating the equilibrium and coordination inherent in the body's kinetic activities.
Stance Phase | 3 months
  Refers to the portion of the gait cycle during which a foot is in contact with the ground. It begins with the initial contact (heel strike) and ends when the same foot leaves the ground (toe-off). The stance phase is a critical component of walking and running, contributing to balance, propulsion, and weight-bearing.
  Measured as a percentage of the total gait cycle, 60% of the cycle in typical walking.
Swing Phase | 3 months
  Refers to the portion of the gait cycle during which a foot is not in contact with the ground. It begins when the foot lifts off the ground (toe-off) and ends when the same foot makes contact again (heel strike). The swing phase allows the leg to advance forward and position itself for the next step. Measured as a percentage of the total gait cycle, 40% of the cycle in normal walking.
Gait Quality Index | 3 months
  The stance-swing phase ratio
First Double support phase | 3 months
  Refers to the portion of the gait cycle during walking when both feet are in contact with the ground simultaneously. It occurs at the beginning of the stance phase for one leg, immediately after heel strike, and ends when the opposite foot lifts off (toe-off). This phase contributes to stability during gait. Measured as a percentage of the total gait cycle.
Single Support Phase | 3 months
  Refers to the portion of the gait cycle during which only one foot is in contact with the ground bearing the entire body weight while the other foot is in the swing phase. It is essential for maintaining balance and forward progression during walking. Measured as a percentage of the total gait cycle.
Propulsion Index | 3 months
  This measures the subject's ability to propel the centre of mass forward during the single support stance phase.
Pelvic tilt range | 3 months
  Refers to the total angular movement of the pelvis in the sagittal plane during a specific activity, such as walking. It represents the difference between the maximum anterior tilt (forward rotation) and maximum posterior tilt (backward rotation) of the pelvis within a given cycle. Measured in degrees (°) to quantify the extent of pelvic rotation.
Pelvic obliquity range | 3 months
  Refers to the total angular movement of the pelvis in the coronal (frontal) plane during activities such as walking. It describes the difference between the maximum upward tilt (hip hike) and maximum downward tilt (hip drop) of one side of the pelvis relative to the opposite side. Measured in degrees (°) to quantify the range of motion.
Pelvic rotation range | 3 months
  Refers to the total angular movement of the pelvis in the transverse (horizontal) plane during activities such as walking. It represents the difference between the maximum forward rotation and maximum backward rotation of the pelvis around a vertical axis within a given cycle. Measured in degrees (°) to quantify the range of rotational motion.
Pelvic symmetry tilt index | 3 months
  Is a quantitative measure that evaluates the symmetry of pelvic tilt during movement. It assesses the degree of deviation in pelvic tilt between the left and right sides in the sagittal plane, providing insight into potential imbalances or asymmetries. Expressed as a percentage (%) to indicate the level of symmetry.
Pelvic symmetry obliquity index | 3 months
  Is a quantitative measure used to evaluate the symmetry of pelvic obliquity during movement. It quantifies the degree of deviation in upward or downward tilt of the pelvis on one side compared to the other in the coronal (frontal) plane, helping to identify potential imbalances or asymmetries. Expressed as a percentage (%) to represent the level of symmetry.
Pelvic symmetry rotation index | 3 months
  Is a quantitative measure used to assess the symmetry of pelvic rotation during movement, particularly in the transverse (horizontal) plane. It calculates the difference in rotational movement between the left and right sides of the pelvis, helping to identify any imbalances or asymmetries in pelvic motion during activities like walking.Expressed as a percentage (%) to indicate the level of symmetry.

SECONDARY OUTCOMES:
Bone remmant (%) | 3 months
  Bone remment respect a healthy femur in percentage (%)
Long discrepancy (mm) | 3 months
  Long discrepancy in milimeters (mm) between healthy and tumoral leg. Positive discrepancy (tumoral leg longer) or negative discrepancy (tumoral leg shorter).

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO LISÓN, PhD, Study Director — Cardenal Herrera University
Locations (1):
- Universidad Ceu Cardenal Herrera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson PJ, Steadman P, Beckman EM, Connick MJ, Carty CP, Tweedy SM. Fitness, Function, and Exercise Training Responses after Limb Salvage With a Lower Limb Megaprosthesis: A Systematic Review. PM R. 2019 May;11(5):533-547. doi: 10.1002/pmrj.12045. Epub 2019 Mar 7. PMID 30844129
- [Background] Morri M, Forni C, Ruisi R, Giamboi T, Giacomella F, Donati DM, Benedetti MG. Postoperative function recovery in patients with endoprosthetic knee replacement for bone tumour: an observational study. BMC Musculoskelet Disord. 2018 Oct 2;19(1):353. doi: 10.1186/s12891-018-2280-7. PMID 30285683